CLINICAL TRIAL: NCT04400032
Title: Cellular Immuno-Therapy for COVID-19 ARDS (CIRCA-19)
Brief Title: Cellular Immuno-Therapy for COVID-19 Acute Respiratory Distress Syndrome
Acronym: CIRCA-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Stem Cell Network (Other); Ontario Research Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20200243-01H
Record Dates: First submitted 2020-04-27; First posted 2020-05-22 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Acute Respiratory Distress Syndrome; Covid19
Keywords: ARDS; COVID-19; Mesenchymal Stromal Cells
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: CIRCA-1901 is is a dose-escalating and safety trial using a 3+3+3 design to determine the safety, and maximum feasible tolerated dose (MFTD) of intravenously (IV) delivered umbilical cord derived MSCs (UC-MSCs). If no safety issues are identified, we will continue to the Phase 2a trial.
  CIRCA-1902 is a single-arm, open-label extension of the CIRCA-1901 trial to assess early signs of efficacy (major morbidity and mortality). The Phase 2a trial (CIRCA-1902) will enroll 12 patients to assess early signals of benefit on mortality and major morbidity in a high risk, high mortality population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Panel 1 (Experimental): 25 million cells/unit dose (cumulative dose: 75 million MSCs)
  Interventions: Biological: Mesenchymal Stromal Cells
- Panel 2 (Experimental): 50 million cells/unit dose (cumulative dose: 150 million MSCs)
  Interventions: Biological: Mesenchymal Stromal Cells
- Panel 3 (Experimental): up to 90 million cells/unit dose (cumulative dose: up to 270 million MSCs)
  Interventions: Biological: Mesenchymal Stromal Cells

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells — The Mesenchymal Stromal Cells will be administered intravenously

SUMMARY:
The clinical picture of the novel corona virus 2 (SARS-CoV-2) disease (COVID-19) is rapidly evolving. Although infections may be mild, up to 25% of all patients admitted to hospital require admission to the intensive care unit, and as many as 40% will progress to develop severe problems breathing due to the acute respiratory distress syndrome (ARDS). ARDS often requires mechanical ventilation, with a 50% risk of mortality. Researchers at the Ottawa Hospital Research Institute (OHRI) have been studying the potential therapeutic role of mesenchymal stromal/stem cells, or MSCs, for the treatment of ARDS for over a decade. This has led to the world's first clinical trial using MSC therapy for patients with severe infections (sepsis) which is often associated with ARDS (NCT02421484). This trial demonstrated tolerability, and potential signs of efficacy. In addition, the investigators have established expertise in producing clinical-grade MSCs and have received approval from Health Canada for the use of MSCs in three different clinical studies.

This protocol consists of 2 sequential trials using the same trial infrastructure, noted as the Phase 1 trial 'CIRCA-1901' and the Phase 2a trial 'CIRCA-1902'. CIRCA-1901 is an open-label, dose-escalating and safety trial using a 3+3+3 design to determine the safety, and maximum feasible tolerated dose of repeated delivery of Umbilical Cord Mesenchymal Stromal Cells (UC-MSC) intravenously. The investigators will enroll up to 9 patients; each receiving repeated unit doses of UC-MSCs delivered by IV infusion on each of 3 consecutive days (24±4 hours apart) according to the following dose-escalation schedule (3 patients per dose panel): (i) Panel 1: 25 million cells/unit dose (cumulative dose: 75 million MSCs), (ii) Panel 2: 50 million cells/unit dose (cumulative dose: 150 million MSCs), (iii) Panel 3: up to 90 million cells/unit dose (cumulative dose: up to 270 million MSCs). If no safety issues are identified, we will continue to the Phase 2a trial.

CIRCA-1902 is a single-arm, open-label extension of the CIRCA-1901 trial to assess early signs of efficacy (major morbidity and mortality). The Phase 2a trial (CIRCA-1902) will enroll 12 patients to assess early signals of benefit on mortality and major morbidity in a high risk, high mortality population.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥18 years
* Laboratory-confirmed SARS-CoV-2 infection during the current admission
* On invasive, non-invasive mechanical ventilation (NIV) (PEEP≥5 cmH20) or high-flow nasal canula (HFNC) oxygen therapy (minimum total flow rate of 40 lpm)
* ARDS (onset <96h) as per the international consensus definition (P/F) ratio < 300 on fraction of inspired oxygen (FiO2)≥0.5, with PEEP ≥5cm H2O or on HFNC), not due to cardiac causes.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this trial:

* No consent/inability to obtain consent
* Moribund patient not expected to survive 24 hours
* Any other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
* Currently receiving extracorporeal life support
* Pregnant or lactating
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Moderate to severe chronic liver disease (Childs-Pugh Score > 12)
* Severe chronic respiratory disease with a baseline PaCO2 > 50 mm Hg or the use of home oxygen
* Lung transplant patient
* Documented deep venous thrombosis or pulmonary embolism within the past 3 months
* Inability/contra-indications to receiving local standard of care thromboprophylaxis
* Chronic immunosuppression (any chronic immunotherapy including daily oral steroid use >6months)
* Known HIV, Hep B/C positive, or active Tuberculosis
* Multisystem shock (SOFA score of >2 in >2 systems)
* Patient, surrogate, or physician not committed to full support including intubation (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | At time of infusion until one year post-infusion
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 to determine the maximum feasible tolerated dose (MFTD) of UC-MSCs given to patients with COVID-19

SECONDARY OUTCOMES:
Number of Participants alive by Day 28 | Day 28
  Number of Participants alive by Day 28
Number of Participants with ventilator-free Days by Day 28 | Day 28
  Number of Participants with ventilator-free Days by Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Duncan J Stewart, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No